CLINICAL TRIAL: NCT00370448
Title: Evaluation of Interventions to Prevent Suicide of Medical Students Through the School-Based Social Support System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CMB-57
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-11

CONDITIONS: Healthy

ARMS (3):
- 1 (Experimental): Training gatekeeper recruited from students and tutors and counselors
  Interventions: Behavioral: school-based social support system
- 2 (Active Comparator)
  Interventions: Behavioral: school-based social support system
- 3 (No Intervention)
  Interventions: Behavioral: school-based social support system

INTERVENTIONS:
Behavioral: school-based social support system — Training gatekeeper recruited from students and tutors and counselors for group 1; training counsellors for group 2; No special intervention for group 3

SUMMARY:
The purpose of this study is to determine whether school-based social support systems are effective in preventing suicide in medical students.

ELIGIBILITY:
Inclusion Criteria:

* Medical university students Grades 1 through 2

Exclusion Criteria:

* Psychopath

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2007-09; Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Rate of suicide ideation | half of one year and one year after intervention

SECONDARY OUTCOMES:
Rate of suicide attempt | half of one year and one year after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yehuan Sun, Ph.D., Study Chair — Anhui Medical University
Locations (1):
- Wannan Medical College, Wuhu, Anhui, China